CLINICAL TRIAL: NCT03571997
Title: FPLLA-PETHEMA-001: Study of Prognostic Factors in Adult Lymphoblastic Lymphoma
Brief Title: Study of Prognostic Factors in Adult Lymphoblastic Lymphoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: PETHEMA Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: FPLLA-PETHEMA-001
Record Dates: First submitted 2018-06-18; First posted 2018-06-28 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Lymphoblastic Lymphoma
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Retrospective observational study with systematic collection of data on filiation (age at diagnosis and sex), clinical data (IPI, ECOG, early response to chemotherapy, overall response to chemotherapy), biological (strain B or T, infiltration of the nervous system central [CNS], bone marrow [MO], lactate dehydrogenase (LDH) level at the time of diagnosis, as well as genetic patients included in the study, as well as the PETHEMA protocol used in the treatment of same patients The study will review the PETHEMA protocols from 2003 to the present

DETAILED DESCRIPTION:
Retrospective observational study with systematic collection of data on filiation (age at diagnosis and sex), clinical data (IPI, ECOG, early response to chemotherapy, overall response to chemotherapy), biological (strain B or T, infiltration of the nervous system central [CNS], bone marrow [MO], lactate dehydrogenase (LDH) level at the time of diagnosis, as well as genetic patients included in the study, as well as the PETHEMA protocol used in the treatment of same patients The study will review the PETHEMA protocols from 2003 to the present. Analysis of the main clinical-biological variables as independent risk factors in adult patients (> 15 years) diagnosed with ALL

ELIGIBILITY:
Inclusion Criteria:

Patients >15 years old diagnosed with ALL and treated with the PETHEMA protocols for ALL

Exclusion Criteria:

None

Min Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients> 15 years diagnosed with ALL and treated with the PETHEMA protocols for ALL
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2018-06-15 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Description pronostic factors | 1 year
  Study of the main clinical-biological variables as independent risk factors in adult patients (> 15 years) diagnosed with ALL

SECONDARY OUTCOMES:
overall survival | 1 year
  To study if there has been an increase in overall survival (OS), in patients diagnosed with ALL in the different PETHEMA protocols
Progression free survival | 1 year
  To study if there has been an increase in progression-free survival (PFS) in patients diagnosed with ALL in the different PETHEMA protocols

CONTACTS AND LOCATIONS:
Locations (28):
- Spain (28):
  - Hospital Mútua de Terrassa, Terrassa, Barcelona
  - Hospital Central de Asturias, Oviedo, Principality of Asturias
  - Hospital General de Alicante, Alicante
  - H. de la Santa Creu I Sant Pau, Barcelona
  - H. Vall d'Hebron, Barcelona, Barcelona
  - H.Universitari Germans Trias I Pujol de Badalona, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital de Basurto, Basurto
  - ICO-Duran i Reynals, Bellvitge
  - Hospital Donostia, Donostia / San Sebastian
  - H. Univ. de Girona Dr. Josep Trueta (ICO), Girona
  - Hospital Arnau de Vilanova (Lleida), Lleida
  - Hospital Lucus Augusti, Lugo
  - H. Gregorio Marañón, Madrid
  - Hospital San Pedro de Alcántara., Málaga
  - Hospital General Universitario Morales Messeguer, Murcia
  - Hospital Son Espases, Palma de Mallorca
  - Hospital Son Llatzer, Palma de Mallorca
  - Complejo Hospitalario de Navarra, Pamplona
  - Parc Taulí, Sabadell
  - H. Univ. de Salamanca, Salamanca
  - C. H. U. de Santiago, Santiago de Compostela
  - Complejo Hosp. Regional Virgen del Rocío, Seville
  - Hospital del Valme, Seville
  - H. Joan XXIII, Tarragona
  - Hoapital La Fe, Valencia
  - Hospital Arnau de Vilanova (Valencia), Valencia
  - Hospital Universitari Clínic València, Valencia

IPD SHARING:
Plan to Share IPD: Undecided